CLINICAL TRIAL: NCT02083406
Title: Open Label Study to Investigate the Pharmacokinetics of Prototype Formulations of OZ439 Administered With Piperaquine Phosphate in the Fasted State to Healthy Subjects
Brief Title: Bioavailability Study of Oral OZ439 Prototype Formulations Administered With Piperaquine Phosphate (PQP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMV_OZ439_13_007
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Malaria
Keywords: Malaria; Bio-availability
MeSH Terms: conditions — Malaria | interventions — Powders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A: OZ439 Prototype 1 (Experimental): 800mg OZ439 prototype formulation 1 and 960mg PQP single doses
  Interventions: Drug: 800mg OZ439 prototype formulation 1; Drug: 960mg PQP
- Treatment B: OZ439 Prototype 2 (Experimental): 800mg OZ439 prototype formulation 2 and 960mg PQP single doses
  Interventions: Drug: 800mg OZ439 prototype formulation 2; Drug: 960mg PQP
- Treatment C: OZ439 Prototype 3 (Experimental): 800mg OZ439 prototype formulation 3 and 960mg PQP single doses
  Interventions: Drug: 800mg OZ439 prototype formulation 3; Drug: 960mg PQP

INTERVENTIONS:
Drug: 800mg OZ439 prototype formulation 1
  Other Names: Treatment A
  Arms: Treatment A: OZ439 Prototype 1
Drug: 800mg OZ439 prototype formulation 2
  Other Names: Treatment B
  Arms: Treatment B: OZ439 Prototype 2
Drug: 800mg OZ439 prototype formulation 3
  Other Names: Treatment C
  Arms: Treatment C: OZ439 Prototype 3
Drug: 960mg PQP
  Other Names: Piperqauine phosphate as powder in bottle

SUMMARY:
A single dose study to investigate how different formulations of OZ439 co-administered with PQP tablest are processed by the body when taken without food

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males, or healthy females of non-childbearing potential ie surgically sterilised or post-menopausal (amenorrhoea for at least 1 year and confirmed by a follicle stimulating hormone result of ≥25 IU/mL
2. Age 18 to 55 years of age
3. Body mass index of 18.0 to 30.0 kg/m2 inclusive. Total body weight >50 kg at screening
4. Willing and able to communicate and participate in the whole study
5. Must provide written informed consent
6. Must agree to use an adequate method of contraception
7. Must have liver function tests and haemoglobin within the laboratory reference range at screening and Day -1
8. Must have heart trace measurements within the defined healthy limits at screening, Day -1 and pre-dose

Exclusion Criteria:

1. Male subjects who have currently pregnant partners
2. Evidence or history of clinically significant oncological, pulmonary, chronic respiratory, hepatic, cardiovascular, haematological, metabolic, neurological, immunological, nephrological, endocrine or psychiatric disease, or current infection
3. Clinically relevant abnormalities in the heart trace including any degree of heart block, including asymptomatic bundle branch block
4. Family history of sudden death or of congenital prolongation of the QTc interval or known congenital prolongation of the QTc interval or any clinical condition known to prolong the QTc interval
5. History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia
6. Electrolyte disturbances, particularly hypokalemia, hypocalcaemia or hypomagnesaemia.
7. Any condition that could possibly affect drug absorption, such as gastrectomy or diarrhoea
8. History of post-antibiotic colitis
9. History of any drug or alcohol abuse in the past 2 years prior to screening
10. Subjects who have a breath carbon monoxide reading of greater than 10 ppm at screening will be excluded. Subjects who are tobacco users (including smokers and users of snuff, chewing tobacco and other nicotine or nicotine-containing products) must have stopped use within 90 days before screening.
11. Receipt of an investigational drug or participation in another clinical research study within 90 days prior to drug administration.
12. Subjects who are study site employees, or immediate family members of a study site or sponsor employee.
13. Subjects who have previously been enrolled in this study
14. Use of ANY prescription or non-prescription medications, vitamins, herbal supplements or dietary supplements, including protein supplements, within 14 days prior to the first dose of study drug and throughout the study, unless prior approval is granted by both the investigator and the sponsor. An exception will be made for intermittent use of paracetamol and hormone replacement therapy. Paracetamol at doses of, at most, 2 g per day or no more than 3 consecutive days or 6 non consecutive days, are allowed until 24 hours before dosing with study drug. Longer exclusion periods apply for:

    1. amiodarone and hydroxychloroquine (210 days)
    2. monoclonal antibodies/ immunoglobulins/ other therapeutic proteins and experimental drugs for which the half-life is not known to the investigator (120 days)
    3. experimental drugs for which half-life is known to the investigator (5 half lives plus 14 days)
    4. chloroquine, piperaquine phosphate and flunarizine (100 days)
    5. fluoxetine (75 days)
    6. benzodiazepines (for midazolam, lorazepam and triazolam, the exclusion period is 14 days), chlorpromazine, mephenytoin, nortryptyline, phenobarbital, primidone, phenprocoumone and cytochrome P450 3A4 inducers not already mentioned, including but not restricted to, rifampin, carbamazepine, oxcarbazepine, phenytoin and St John's Wort (35 days)
15. Positive hepatitis B surface antigen, hepatitis C virus antibody or human immunodeficiency virus results
16. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator
17. Positive urine drug screen result at screening or admission to the clinical unit
18. History of intolerance or hypersensitivity to piperaquine or any 4-aminoquinolone, or ascertained or presumptive hypersensitivity to the active principle and/or formulation ingredients; history of anaphylaxis to drugs or allergic reactions in general, that the investigator considers may affect the outcome of the study
19. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
20. Presence or history of allergy requiring treatment; hayfever is allowed unless it is active
21. Donation or loss of >400 mL of blood within 90 days prior to drug administration
22. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
23. Subjects who do not have suitable veins for multiple blood samples as assessed by the investigator at screening
24. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jo Collier, MBChB FFPM, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Nottingham, Nottinghamshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A: OZ439 Prototype 1: 800mg OZ439 prototype formulation 1 and 960mg PQP single doses under fasted conditions
- Treatment B: OZ439 Prototype 2: 800mg OZ439 prototype formulation 2 and 960mg PQP single doses under fasted conditions
- Treatment C: OZ439 Prototype 3: 800mg OZ439 prototype formulation 3 and 960mg PQP single doses under fasted conditions
Period: Overall Study
Arm/Group | Treatment A: OZ439 Prototype 1 | Treatment B: OZ439 Prototype 2 | Treatment C: OZ439 Prototype 3
Started | 7 | 8 | 7
Completed | 7 | 8 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A: OZ439 Prototype 1 | Treatment B: OZ439 Prototype 2 | Treatment C: OZ439 Prototype 3 | Total
Number analyzed (Participants) | 7 | 8 | 7 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (8.2) | 44.9 (11.3) | 35.7 (4.1) | 36.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 0 | 2
  Male | 7 | 6 | 7 | 20
Region of Enrollment [Number; unit: participants]
  United Kingdom | 7 | 8 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: OZ439 AUC(0-168h)
Description: OZ439 Area under the plasma concentration (AUC) versus time curve
Time Frame: Up to 168 hours post-dose
Population: All subjects who received at least one dose of study drug and had sufficient plasma concentration data for pharmacokinetics (PK) parameter estimation
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: OZ439 Prototype 1 | Treatment B: OZ439 Prototype 2 | Treatment C: OZ439 Prototype 3
Number analyzed (Participants) | 7 | 8 | 7
ng*h/mL | 8780 (43.7) | 10300 (23.7) | 9460 (43.0)

2. Primary Outcome: OZ439 Cmax
Description: OZ439 Maximum observed concentration
Time Frame: Up to 168 hours post-dose
Population: All subjects who received at least one dose of study drug and had sufficient plasma concentration data for PK parameter estimation
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: OZ439 Prototype 1 | Treatment B: OZ439 Prototype 2 | Treatment C: OZ439 Prototype 3
Number analyzed (Participants) | 7 | 8 | 7
ng/mL | 877 (41.3) | 995 (32.2) | 924 (50.5)

3. Secondary Outcome: Piperaquine (PQ) AUC(0-168h)
Description: PQ Area under the plasma concentration versus time curve
Time Frame: Up to 168h post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: OZ439 Prototype 1 | Treatment B: OZ439 Prototype 2 | Treatment C: OZ439 Prototype 3
Number analyzed (Participants) | 7 | 8 | 7
ng*h/mL | 3730 (41.3) | 2810 (21.8) | 3300 (50.7)

4. Secondary Outcome: PQ Cmax
Description: PQ Maximum observed concentration
Time Frame: Up to 168h post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: OZ439 Prototype 1 | Treatment B: OZ439 Prototype 2 | Treatment C: OZ439 Prototype 3
Number analyzed (Participants) | 7 | 8 | 7
ng/mL | 99.8 (90.1) | 89.5 (54.1) | 91.2 (130.8)

ADVERSE EVENTS:
Time Frame: Up to Day 43 post-dose
Description: All 22 subjects received one dose of OZ439 in combination with PQP and were included in the safety analysis population
Arm/Group | Treatment A: OZ439 Prototype 1 | Treatment B: OZ439 Prototype 2 | Treatment C: OZ439 Prototype 3
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 2/7 | 7/8 | 2/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: OZ439 Prototype 1 (N=7) | Treatment B: OZ439 Prototype 2 (N=8) | Treatment C: OZ439 Prototype 3 (N=7)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No